CLINICAL TRIAL: NCT03284099
Title: Is Bedtime Administration of ACEIs and ARBs More Effective for Reverting Non-dipper Status Than Morning Administration for Non-dipping Hypertension in Hong Kong Primary Care? A Pilot Study
Brief Title: Bedtime ACEIs/ARBs Versus Morning ACEIs/ARBs for Reverting Non-dipping Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding obtained. The ABPM machines are being used for another project
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.182-T
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Hypertension; Non-Dipping
MeSH Terms: conditions — Hypertension | interventions — Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): ACEIs or ARBs will be switch to be taken before bedtime
  Interventions: Drug: ACEi, ARB
- control (Active Comparator): ACEIs or ARBs will be taken in the morning as usual
  Interventions: Drug: ACEi, ARB

INTERVENTIONS:
Drug: ACEi, ARB — To take the ACEis or ARBs before bedtime instead of in the morning

SUMMARY:
Background: Non-dipping (ND), defined as a <10% decrease in blood pressure (BP) during sleep, is an independent significant predictor of cardiovascular outcome in hypertensive patients. A few anti-hypertensive medications, including angiotensin receptor blockers (ARBs) and angiotensin converting enzyme inhibitors (ACEIs), may normalize dipping if administered at night. Chinese data are scarce and there are no prospective studies on cardiovascular outcomes in Chinese patients.

Aim: To determine if the bedtime administration of ACEIs and ARBs is more effective at normalizing ND than morning administration. As a pilot project, the feasibility of recruiting hypertension patients in primary care for ambulatory blood pressure monitoring (ABPM) and conducting a clinical trial will be evaluated such that future larger randomized trials can be planned to determine treatments for ND.

Method: Fifty patients diagnosed with essential hypertension who are receiving either ACEIs or ARBs and diagnosed with ND will be randomized to take ACEIs or ARBs either early morning or before bedtime. A follow-up 48-hour ABPM will be performed after 4-6 weeks to examine post-treatment changes in BP and ND status.

Outcome: The primary outcome of this proposed study is the proportion of ND at 6 weeks; secondary outcomes will include (i) mean awake and asleep SBP/DBP of 48-hour duration (ii) feasibility of this pilot study will be assessed by recruitment and dropout rates during the study period.

Potential: This pilot study will provide the basis for a future larger randomized controlled study to further examine the treatment for ND in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are taking an ACEI or an ARB
* >18 years of age
* Chinese and
* Received a diagnosis of primary HT.

Exclusion Criteria:

* Severe HT as defined by a clinic systolic BP ≥180 mmHg and/or diastolic BP ≥ 110 mmHg
* allergic reaction or intolerance to the current ACEI or ARB
* unable to provide consent
* pregnancy
* night-time worker
* occupational drivers since patients will be asked not to move during BP measurements, which may induce potential danger in driving
* taking anti-coagulants to avoid causing bruises when using ABPM
* known atrial fibrillation since ABPM use has not been validated in this group
* known hyperkalemia
* ABPM discovered hypotension (mean SBP < 100 and/or mean DBP < 60) because these patients may need to stop their medications
* Reported sleep time of <4 hours per night (at least seven readings are recommended during sleep for an ABPM recording to be valid, and a sleeping time < 4 hours is unlikely to generate valid results).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of non-dipping in each group as measured by ambulatory BP machines(ABPM) | 6 weeks
  the ABPM - An ApneABP (Meditech, Hungary) will be used in the study. non-dipping is defined as lack of more than 10% drop in SBP during sleep when compared to awake BP. The sleep duration and time are defined by actigraphy (Actigraph, model GT9X-BT)

SECONDARY OUTCOMES:
mean awake and asleep SBP/DBP of 48-hour duration as assessed by ABPM | 6 weeks
feasibility of the intervention as assessed by dropout rate | 1 year (assessed after the whole study)
  The trial is deemed feasible and a larger similar study can be conducted if: (i) ≤30% of ND patients drop out from the study

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
to decide after end of trial